CLINICAL TRIAL: NCT02216045
Title: Investigating the Effects of Camel Milk Products on the Laboratory Markers in the Patients With Chronic Hepatitis C, Genotype 2 & 3
Brief Title: Effect of Camel Milk on Chronic Hepatitis C
Acronym: HCV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, mohammadreza noras, Phd student, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mashhad UMS
Record Dates: First submitted 2014-07-26; First posted 2014-08-13 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C ,Chronic Hepatitis C ,camel milk
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peginterferon ,Ribavirin (Active Comparator): drug :Peginterferon, Ribavirin,
  Interventions: Drug: Peginterferon, Ribavirin
- Peginterferon, Ribavirin, camel milk (Experimental): drug :Peginterferon, Ribavirin, camel milk
  Interventions: Drug: Peginterferon, Ribavirin, camel milk

INTERVENTIONS:
Drug: Peginterferon, Ribavirin, camel milk — Peginterferon One subcutaneous injection containing 0.5 ml solution with180 mcg PegIFNα-2a per week for 12 weeks.
  Ribavirin (RBV) tablets (body-weight adjusted dose: < 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) taken orally (by mouth) once daily for for 12 weeks .
  camel milk 250 ml of raw camel milk will be consumed in 10 minutes orally twice daily for 12 weeks.
  Other Names: PEGASYS® COPEGUS®. Dromedary milk (camel milk )
  Arms: Peginterferon, Ribavirin, camel milk
Drug: Peginterferon, Ribavirin — Peginterferon (PegIFNα-2a) One subcutaneous injection containing 0.5 ml solution with180 mcg PegIFNα-2a per week for 12 weeks.
  Ribavirin (RBV) tablets (body-weight adjusted dose: < 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) taken orally (by mouth) once daily for for 12 weeks.
  Other Names: PEGASYS® (Peginterferon ) , COPEGUS® (Ribavirin)
  Arms: Peginterferon ,Ribavirin

SUMMARY:
Camel milk as the new modality for treatment of chronic hepatitis C. The purpose of this study is to evaluate effectiveness and safety of camel milk in combination with Peginterferon Alfa-2a and Ribavirin in genotype 2,3 chronic hepatitis C virus .

DETAILED DESCRIPTION:
The investigators enrolled 40 patients into the study. Group 1(Intervention ) : received PEGASYS( Peginterferon ) One subcutaneous injection containing 0.5 ml solution with180 mcg per week plus COPEGUS( Ribavirin ) tablets (body-weight adjusted dose: < 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) taken orally (by mouth) once daily and 250 ml of raw camel milk will be consumed in 10 minutes orally twice daily for 12 weeks.

Group 2 ( control ): received PEGASYS( Peginterferon ) One subcutaneous injection containing 0.5 ml solution with180 mcg per week plus COPEGUS( Ribavirin ) tablets (body-weight adjusted dose: < 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) taken orally (by mouth) once daily for 12 weeks.

Follow up period is 1,2,3 months after treatment. The patients are visited every 4 weeks with biochemistry lab tests. The patients are checked with quantitative HCV RNA (Ribonucleic Acid) on the first months after initiation of the treatment to assess early virologic response and at the end of the study for complete response rate and on the third month after treatment completion for sustained response rate. The patients with undetectable HCV RNA are considered as responders.

ELIGIBILITY:
Inclusion Criteria:

* HCV (hepatitis C virus ) RNA positive
* Age age groups (18 to 70 years)

Exclusion Criteria:

* Ongoing pregnancy or breast feeding
* Hx of HCC(hepatocellular carcinoma )
* Hx of alcoholic liver disease
* Hx of bleeding from esophageal varices
* Hx of hemochromatosis
* Hx of autoimmune hepatitis
* Hx of Suicidal attempt
* Hx of cerebrovascular dis
* Hx of severe retinopathy
* Hx of severe psoriasis
* Hx of scleroderma
* Hx of metabolic liver disease
* Hx of SLE(systemic lupus erythematosus )

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Early Virologic Responses(EVR) | After 4 weeks of Treatment
  Change From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (log10 IU/mL) at Week 4 in Treatment by PEG IFN ( interferon) + RBV.
Early Virologic Responses(EVR) | 4 weeks after of treatment
  Change From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (log10 IU/mL) at Week 4 in Treatment by PEG IFN + RBV+camel milk

SECONDARY OUTCOMES:
Complete early virological response (cEVR) | 12 weeks after initiation of treatment
  defined by undetectable HCV RNA at 12 weeks post initiation of dual therapy by PEG IFN + RBV
o Complete early virological response (cEVR) | 12 weeks after initiation of treatment
  defined by undetectable HCV RNA at 12 weeks post initiation of dual therapy by PEG IFN + RBV+camel milk
o Sustained virological response (SVR) | 12 weeks after initiation of treatment
  defined by HCV RNA below the detection limit based on quantitative PCR 12 weeks after stopping treatment by PEG IFN +RBV
o Sustained virological response (SVR) | 12 weeks after initiation of treatment
  defined by HCV RNA below the detection limit based on quantitative PCR(polymerase chain reaction ) 12 weeks after stopping treatment by PEG IFN +RBV+camel milk
o Normalization of ALT( Alanine Aminotransferase) | during the treatment and 12 weeks of treatment
  Proportion of patients who have ALT below the upper limit of normal (ULN) during the treatment by PEG IFN +RBV and 12 weeks after the end of treatment.
o Normalization of ALT | during the treatment and 12 weeks of treatment
  Proportion of patients who have ALT below the upper limit of normal (ULN) during the treatment by PEG IFN +RBV+camel milk and 12 weeks after of treatment.
o Adverse events(AE) | Up to 12 weeks
  Number of participants experiencing adverse events
o Adverse events(AE) | Up to 12 weeks
  Number of participants discontinuing study treatment because of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Seyyd Musa Al-Reza Hosseini, professor.As, Study Chair — Ghaem Gastrointestinal Clinic; Mehdi Yousefi, MD.Phd, Study Director — Faculty of Traditional Medicine Clinic; Mohammadreza Noras, Phd student, Principal Investigator — Faculty of Traditional Medicine Clinic; Ali Taghipour, MD.Phd, Study Director — MUMS Faculty of Health Sciences; Said Zibae, MD.Phd, Study Director — Razi vaccine and serum Research Institue of Mashhd
Locations (2):
- Iran (2):
  - Faculty of Traditional Medicine, Mashhad, Razavi Khorasan Province
  - Mashhad University of Medical Sciences, Mashhad, Razavi Khorasan Province

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) is confidential in researchers .